CLINICAL TRIAL: NCT04868630
Title: Calibration of the Average Breathing Rate Measurement of the Cloud DX Pulsewave Health Monitor (PAD-2A) Device (CCV-3)
Acronym: CCV-3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardiovascular Research New Brunswick (Other)
Collaborators: Cloud DX Inc. (Industry); Horizon Health Network (Other); Atlantic Sleep Center (Unknown); New Brunswick Health Research Foundation (Other); Dalhousie University (Other)
Responsible Party: Sponsor
Other Study IDs: RS#: 2020-2908; R#: 100948; STP-PW2-001 (Other: Health Canada)
Record Dates: First submitted 2021-04-21; First posted 2021-05-03 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Outpatients
Keywords: average breathing rate (breath per minute); vital sign monitoring; telemedicine; non-invasive device

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Outpatients; Atlantic Sleep Centre & SJRH Respiratory Clinic: The study population consists of approximately 80 adult, outpatient participants recruited from the Atlantic Sleep Centre and the Respiratory Clinic at the Horizon Health Network, Saint John Regional Hospital.
  Interventions: Device: Pulsewave Health Monitor (PAD-2A) Device

INTERVENTIONS:
Device: Pulsewave Health Monitor (PAD-2A) Device — This is an observational study of the average breathing rate measurement of a non-invasive wrist cuff device. The purpose of this study is to calibrate the average breathing rate measurement of the Pulsewave Health Monitor (PAD-2A) wrist cuff device with the breathing rate measurement of a standard clinical capnography device. Additionally, we will also compare the average breathing rate measurement of the capnography device with other standard clinical respiratory devices (i.e. nasal pressure transducer, thermistor, and respiratory inductance plethysmography (RIP) belts of the chest and abdomen).

SUMMARY:
The purpose of this study is to calibrate the average breathing rate measurement of the PAD-2A device to be within ±2 breaths per minute of clinical capnography breathing rate measurements.

DETAILED DESCRIPTION:
The plan for this study is to calibrate the average breathing rate measurement of the PAD-2A device with the breathing rate measurement of a standard clinical capnography device. The data will be collected and analyzed in order to calibrate the PAD-2A device via the capnography measures by adjusting the device algorithm for the breathing rate measurements to be within ±2 breaths per minute. Additionally, the secondary objective of this study is to compare the clinical standard respiratory rate measurement of capnography with the respiratory rate measurements of other standard clinical respiratory devices (i.e. nasal pressure transducer, thermistor, and the respiratory inductance plethysmography (RIP) belts of the chest and abdomen).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 19 years of age (minimum 30% male/female)
* Wrist circumference between 13.5cm - 23cm (5.3 in. - 9.1in.)

  * Specifically for this test device, the wrist size of the consented participants will be distributed accordingly for a Gaussian distribution:

Lowest Octile: ≥ 13.5cm to < 14.7cm Lower Quarter: ≥ 13.5cm to < 15.9cm Lower-Middle Quarter: ≥ 15.9cm to < 18.3cm Upper-Middle Quarter: ≥ 18.3cm to < 20.7cm Upper Quarter: ≥ 20.7cm to ≤ 23.0cm Highest Octile: ≥ 21.9cm to ≤ 23.0cm

• Willing to volunteer to participate and to sign the study specific informed consent form

Exclusion Criteria:

* Wrist circumference less than 13.5cm (5.3 in.) or greater than 23cm (9.1 in)
* Hand or body tremors
* Canadian Cardiovascular Society (CCS) grade III or IV angina pectoris (chest pain)
* Unexplained shortness of breath at rest
* History of seizures (except childhood febrile seizures)
* Epilepsy
* History of unexplained syncope (fainting)
* Pregnant
* A musculoskeletal disorder that prevents a non-invasive device to be inflated/deflated on the arm
* Unwilling to volunteer to participate and to sign the study specific informed consent form

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For the PAD-2A device calibration phase of the study, we will recruit and consent approximately 80 adult male and female patient participants (≥ 19 years of age; minimum 30% male/female) who are referred to the Atlantic Sleep Centre or the Respiratory Clinic at the Saint John Regional Hospital (SJRH) and who are willing to volunteer to participate in the study. Eligibility of participants will be determined based on the inclusion/exclusion criteria of the study, as described below.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Breathing rate | From the start of cuff deflation to the end of cuff deflation (approximately 60 seconds).
  Non-invasive Pulsewave Health Monitor (PAD-2A) wrist cuff device (breaths per minute)
Breathing rate | Simultaneous measurement with the PAD-2A wrist cuff device from the start of cuff deflation to the end of cuff deflation (approximately 60 seconds).
  Standard clinical capnograph device via nasal cannula (breaths per minute)
Breathing rate | Simultaneous measurement with the PAD-2A wrist cuff device from the start of cuff deflation to the end of cuff deflation (approximately 60 seconds).
  Standard clinical nasal pressure transducer via nasal cannula (breaths per minute)
Breathing rate | Simultaneous measurement with the PAD-2A wrist cuff device from the start of cuff deflation to the end of cuff deflation (approximately 60 seconds).
  Standard clinical thermistor via nasal cannula (breaths per minute)

SECONDARY OUTCOMES:
Breathing rate | Simultaneous measurement with the PAD-2A wrist cuff device from the start of cuff deflation to the end of cuff deflation (approximately 60 seconds).
  Standard clinical respiratory inductance plethysmography (RIP) belts (breaths per minute)

CONTACTS AND LOCATIONS:
Overall Officials: Graham Bishop, MD, FRCP(C), Principal Investigator — Atlantic Sleep Centre
Locations (1):
- Horizon Health Network, Saint John, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Currently, the clinical research group is undecided regarding individual participant data (IPD) sharing with other researchers upon completion of this study, although it is acknowledged that the practice of data sharing among scientists, clinicians, and other professionals is of increasing importance, particularly for transparency in clinical research studies.

REFERENCES:
- See also: Cloud DX device company website. — https://clouddx.com/